CLINICAL TRIAL: NCT00006164
Title: Hepatitis C Antiviral Long-term Treatment Against Cirrhosis Trial (HALT-C)
Brief Title: Long Term Interferon for Patients Who Did Not Clear Hepatitis C Virus With Standard Treatment
Acronym: HALT-C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH); National Cancer Institute (NCI) (NIH); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HALT C; N01-DK-9-2328 (Other Grant/Funding Number: NIH NIDDK Contract); N01-DK-9-2323 (Other Grant/Funding Number: NIH NIDDK Contract); N01-DK-9-2324 (Other Grant/Funding Number: NIH NIDDK Contract); N01-DK-9-2325 (Other Grant/Funding Number: NIH NIDDK Contract); N01-DK-9-2326 (Other Grant/Funding Number: NIH NIDDK Contract); N01-DK-9-2321 (Other Grant/Funding Number: NIH NIDDK Contract); N01-DK-9-2327 (Other Grant/Funding Number: NIH NIDDK Contract); N01-DK-9-2319 (Other Grant/Funding Number: NIH NIDDK Contract); N01-DK-9-2318 (Other Grant/Funding Number: NIH NIDDK Contract); N01-DK-9-2320 (Other Grant/Funding Number: NIH NIDDK Contract); N01-DK-9-2322 (Other Grant/Funding Number: NIH NIDDK Contract); NCT00006139 (obsolete NCT alias)
Record Dates: First submitted 2000-08-08; First posted 2000-08-09 (Estimated); Results first posted 2009-09-04 (Estimated); Last update posted 2020-05-12 (Actual); Status verified 2020-04

CONDITIONS: Chronic Hepatitis c; Cirrhosis, Liver; Fibrosis, Liver; Hepatic Cirrhosis
Keywords: liver disease; hepatitis c virus; antiviral agent; cirrhosis
MeSH Terms: conditions — Hepatitis C, Chronic; Liver Cirrhosis; Liver Diseases; Hepatitis C; Fibrosis | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): Peg-interferon alfa-2a 90 mcg/week
  Interventions: Drug: Peginterferon alfa-2a + Ribavirin; Drug: Peginterferon alfa-2a
- 2 (Active Comparator): Standard of care followup
  Interventions: Drug: Peginterferon alfa-2a + Ribavirin

INTERVENTIONS:
Drug: Peginterferon alfa-2a + Ribavirin — Peginterferon alfa-2a 180 mcg/week injection, for 24 weeks, plus 1000-1200 mg Ribavirin oral (prescribed according to weight <75 kg, >75 kg) daily in two divided doses for 24 weeks
  Other Names: Pegasys (Hoffman-La Roche); Copegus (Hoffman-La Roche)
Drug: Peginterferon alfa-2a — 90 mcg/week injection, for 3.5 years
  Other Names: Pegasys (Hoffman-La Roche)
  Arms: 1

SUMMARY:
The HALT-C Trial is a National Institute of Diabetes and Digestive and Kidney Diseases sponsored, randomized clinical trial of long-term use of Peginterferon alfa-2a (pegylated interferon) in patients who failed to respond to prior interferon treatment. All patients who enter the trial will be treated for 6 months with Peginterferon alfa-2a and Ribavirin. Patients who respond to this 6 month treatment will continue to be treated for an additional 6 months.

Patients who do not respond to this treatment will be eligible for the long-term maintenance phase of this study where patients will be randomly selected to be treated with Peginterferon alfa-2a or to discontinue treatment for 3.5 years. Patients in both arms of this study will be followed closely with quarterly study visits.

The combination of peginterferon plus ribavirin has recently been approved by the FDA for treatment of chronic hepatitis C. Patients who remain HCV-RNA positive after being treated for at least 6 months with peginterferon and ribavirin outside of this study may be eligible to directly enter the randomized portion of the HALT-C Trial.

The HALT-C study is designed to determine if continuing interferon long-term over several years will suppress Hepatitis C virus, prevent progression to cirrhosis, prevent liver cancer and reduce the need for liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age at entry at least 18 years.
* Positive for Hepatitis C.
* Previous treatment with any interferon or interferon and ribavirin for at least 3 months.
* Documented non-response to treatment with interferon.
* A liver biopsy demonstrating significant liver scarring.

Exclusion Criteria:

* No other liver disease.
* No unstable major medical diseases or conditions.
* No major complications of cirrhosis.
* No recent abuse of alcohol or illicit drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Actual)
Dates: Start 2000-06 (Actual); Primary Completion 2007-04 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory T. Everson, M.D., Principal Investigator — UCHSC (University of Colorado); Adrian M. Di Bisceglie, M.D., Principal Investigator — St. Louis University; William M. Lee, M.D., Principal Investigator — University of Texas, Southwestern Medical Center at Dallas; Marc Ghany, M.D., Principal Investigator — LDS, NIDDK, NIH; Jules L. Dienstag, M.D., Principal Investigator — Massachusetts General Hospital; Mitchell Shiffman, M.D., Principal Investigator — Medical College of Virginia; Anna Lok, M.D., Principal Investigator — University of Michigan; Tim Morgan, M.D., Principal Investigator — University of California-Irvine/VA Medical Center-Long Beach; Karen Lindsay, M.D., M.M.M., Principal Investigator — USC School of Medicine; Gyongyi Szabo, M.D., Ph.D., Principal Investigator — UMass Medical School
Locations (11):
- United States (11):
  - University of California-Irvine/VA Medical Center-Long Beach, Long Beach, California
  - USC School of Medicine, Los Angeles, California
  - UCHSC (University of Colorado), Denver, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Lds, Niddk, Nih, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - UMass Memorial HealthCare, University Campus, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Saint Louis University, St Louis, Missouri
  - University of Texas Southwestern - Dallas, Dallas, Texas
  - Medical College of Virginia, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Data are available at the NIDDK Central Repository: https://repository.niddk.nih.gov/studies/halt-c/?query=HALT-C
URL: https://repository.niddk.nih.gov/studies/halt-c/?query=HALT-C

REFERENCES:
- [Background] Lee WM, Dienstag JL, Lindsay KL, Lok AS, Bonkovsky HL, Shiffman ML, Everson GT, Di Bisceglie AM, Morgan TR, Ghany MG, Morishima C, Wright EC, Everhart JE; HALT-C Trial Group. Evolution of the HALT-C Trial: pegylated interferon as maintenance therapy for chronic hepatitis C in previous interferon nonresponders. Control Clin Trials. 2004 Oct;25(5):472-92. doi: 10.1016/j.cct.2004.08.003. PMID 15465617
- [Result] Di Bisceglie AM, Shiffman ML, Everson GT, Lindsay KL, Everhart JE, Wright EC, Lee WM, Lok AS, Bonkovsky HL, Morgan TR, Ghany MG, Morishima C, Snow KK, Dienstag JL; HALT-C Trial Investigators. Prolonged therapy of advanced chronic hepatitis C with low-dose peginterferon. N Engl J Med. 2008 Dec 4;359(23):2429-41. doi: 10.1056/NEJMoa0707615. PMID 19052125
- [Derived] Yu L, Paski SC, Dodge J, Bambha K, Biggins SW, Ioannou GN. Effect of dietary branched chain amino acids on liver related mortality: Results from a large cohort of North American patients with advanced HCV infection. PLoS One. 2023 Apr 25;18(4):e0284739. doi: 10.1371/journal.pone.0284739. eCollection 2023. PMID 37098004
- [Derived] Donlin MJ, Lomonosova E, Kiss A, Cheng X, Cao F, Curto TM, Di Bisceglie A, Tavis JE. HCV genome-wide genetic analyses in context of disease progression and hepatocellular carcinoma. PLoS One. 2014 Jul 31;9(7):e103748. doi: 10.1371/journal.pone.0103748. eCollection 2014. PMID 25079603
- [Derived] Snow KK, Bell MC, Stoddard AM, Curto TM, Wright EC, Dienstag JL. Processes to manage analyses and publications in a phase III multicenter randomized clinical trial. Trials. 2014 May 7;15:159. doi: 10.1186/1745-6215-15-159. PMID 24886378
- [Derived] Morishima C, Shiffman ML, Dienstag JL, Lindsay KL, Szabo G, Everson GT, Lok AS, Di Bisceglie AM, Ghany MG, Naishadham D, Morgan TR, Wright EC; HALT-C Trial Group. Reduction in Hepatic Inflammation Is Associated With Less Fibrosis Progression and Fewer Clinical Outcomes in Advanced Hepatitis C. Am J Gastroenterol. 2012 Sep;107(9):1388-98. doi: 10.1038/ajg.2012.137. Epub 2012 Jun 12. PMID 22688849
- [Derived] Morishima C, Di Bisceglie AM, Rothman AL, Bonkovsky HL, Lindsay KL, Lee WM, Koziel MJ, Fontana RJ, Kim HY, Wright EC; HALT-C Trial Group. Antigen-specific T lymphocyte proliferation decreases over time in advanced chronic hepatitis C. J Viral Hepat. 2012 Jun;19(6):404-13. doi: 10.1111/j.1365-2893.2011.01562.x. Epub 2011 Dec 16. PMID 22571902
- [Derived] Fontana RJ, Litman HJ, Dienstag JL, Bonkovsky HL, Su G, Sterling RK, Lok AS; HALT-C Trial Group. YKL-40 genetic polymorphisms and the risk of liver disease progression in patients with advanced fibrosis due to chronic hepatitis C. Liver Int. 2012 Apr;32(4):665-74. doi: 10.1111/j.1478-3231.2011.02686.x. Epub 2011 Nov 22. PMID 22103814
- [Derived] Everson GT, Shiffman ML, Hoefs JC, Morgan TR, Sterling RK, Wagner DA, Lauriski S, Curto TM, Stoddard A, Wright EC; HALT-C Trial Group. Quantitative liver function tests improve the prediction of clinical outcomes in chronic hepatitis C: results from the Hepatitis C Antiviral Long-term Treatment Against Cirrhosis Trial. Hepatology. 2012 Apr;55(4):1019-29. doi: 10.1002/hep.24752. Epub 2012 Mar 1. PMID 22030902
- [Derived] Sterling RK, Wright EC, Morgan TR, Seeff LB, Hoefs JC, Di Bisceglie AM, Dienstag JL, Lok AS. Frequency of elevated hepatocellular carcinoma (HCC) biomarkers in patients with advanced hepatitis C. Am J Gastroenterol. 2012 Jan;107(1):64-74. doi: 10.1038/ajg.2011.312. Epub 2011 Sep 20. PMID 21931376
- [Derived] O'Bryan JM, Potts JA, Bonkovsky HL, Mathew A, Rothman AL; HALT-C Trial Group. Extended interferon-alpha therapy accelerates telomere length loss in human peripheral blood T lymphocytes. PLoS One. 2011;6(8):e20922. doi: 10.1371/journal.pone.0020922. Epub 2011 Aug 4. PMID 21829595
- [Derived] Rakoski MO, Brown MB, Fontana RJ, Bonkovsky HL, Brunt EM, Goodman ZD, Lok AS, Omary MB; HALT-C Trial Group. Mallory-Denk bodies are associated with outcomes and histologic features in patients with chronic hepatitis C. Clin Gastroenterol Hepatol. 2011 Oct;9(10):902-909.e1. doi: 10.1016/j.cgh.2011.07.006. Epub 2011 Jul 23. PMID 21782771
- [Derived] O'Brien TR, Everhart JE, Morgan TR, Lok AS, Chung RT, Shao Y, Shiffman ML, Dotrang M, Sninsky JJ, Bonkovsky HL, Pfeiffer RM; HALT-C Trial Group. An IL28B genotype-based clinical prediction model for treatment of chronic hepatitis C. PLoS One. 2011;6(7):e20904. doi: 10.1371/journal.pone.0020904. Epub 2011 Jul 8. PMID 21760886
- [Derived] Hoefs JC, Shiffman ML, Goodman ZD, Kleiner DE, Dienstag JL, Stoddard AM; HALT-C Trial Group. Rate of progression of hepatic fibrosis in patients with chronic hepatitis C: results from the HALT-C Trial. Gastroenterology. 2011 Sep;141(3):900-908.e1-2. doi: 10.1053/j.gastro.2011.06.007. Epub 2011 Jun 12. PMID 21699796
- [Derived] Dienstag JL, Ghany MG, Morgan TR, Di Bisceglie AM, Bonkovsky HL, Kim HY, Seeff LB, Szabo G, Wright EC, Sterling RK, Everson GT, Lindsay KL, Lee WM, Lok AS, Morishima C, Stoddard AM, Everhart JE; HALT-C Trial Group. A prospective study of the rate of progression in compensated, histologically advanced chronic hepatitis C. Hepatology. 2011 Aug;54(2):396-405. doi: 10.1002/hep.24370. Epub 2011 Jun 23. PMID 21520194
- [Derived] Freedman ND, Curto TM, Lindsay KL, Wright EC, Sinha R, Everhart JE; HALT-C TRIAL GROUP. Coffee consumption is associated with response to peginterferon and ribavirin therapy in patients with chronic hepatitis C. Gastroenterology. 2011 Jun;140(7):1961-9. doi: 10.1053/j.gastro.2011.02.061. Epub 2011 Mar 2. PMID 21376050
- [Derived] Lok AS, Everhart JE, Di Bisceglie AM, Kim HY, Hussain M, Morgan TR; HALT-C Trial Group. Occult and previous hepatitis B virus infection are not associated with hepatocellular carcinoma in United States patients with chronic hepatitis C. Hepatology. 2011 Aug;54(2):434-42. doi: 10.1002/hep.24257. PMID 21374690
- [Derived] Lambrecht RW, Sterling RK, Naishadham D, Stoddard AM, Rogers T, Morishima C, Morgan TR, Bonkovsky HL; HALT-C Trial Group. Iron levels in hepatocytes and portal tract cells predict progression and outcomes of patients with advanced chronic hepatitis C. Gastroenterology. 2011 May;140(5):1490-500.e3. doi: 10.1053/j.gastro.2011.01.053. Epub 2011 Feb 15. PMID 21335007
- [Derived] Fontana RJ, Sanyal AJ, Ghany MG, Bonkovsky HL, Morgan TR, Litman HJ, Reid AE, Lee WM, Naishadham D; HALT-C Trial Study Group. Development and progression of portal hypertensive gastropathy in patients with chronic hepatitis C. Am J Gastroenterol. 2011 May;106(5):884-93. doi: 10.1038/ajg.2010.456. Epub 2010 Dec 7. PMID 21139575
- [Derived] Lok AS, Everhart JE, Wright EC, Di Bisceglie AM, Kim HY, Sterling RK, Everson GT, Lindsay KL, Lee WM, Bonkovsky HL, Dienstag JL, Ghany MG, Morishima C, Morgan TR; HALT-C Trial Group. Maintenance peginterferon therapy and other factors associated with hepatocellular carcinoma in patients with advanced hepatitis C. Gastroenterology. 2011 Mar;140(3):840-9; quiz e12. doi: 10.1053/j.gastro.2010.11.050. Epub 2010 Dec 1. PMID 21129375
- [Derived] Freedman ND, Curto TM, Morishima C, Seeff LB, Goodman ZD, Wright EC, Sinha R, Everhart JE; HALT-C Trial Group. Silymarin use and liver disease progression in the Hepatitis C Antiviral Long-Term Treatment against Cirrhosis trial. Aliment Pharmacol Ther. 2011 Jan;33(1):127-37. doi: 10.1111/j.1365-2036.2010.04503.x. Epub 2010 Nov 2. PMID 21083592
- [Derived] Kronfol Z, Litman HJ, Back-Madruga C, Bieliauskas LA, Lindsay KL, Lok AS, Fontana RJ; HALT-C Trial Group. No increase in depression with low-dose maintenance peginterferon in prior non-responders with chronic hepatitis C. J Affect Disord. 2011 Mar;129(1-3):205-12. doi: 10.1016/j.jad.2010.09.010. PMID 20889211
- [Derived] Fontana RJ, Dienstag JL, Bonkovsky HL, Sterling RK, Naishadham D, Goodman ZD, Lok AS, Wright EC, Su GL; HALT-C Trial Group. Serum fibrosis markers are associated with liver disease progression in non-responder patients with chronic hepatitis C. Gut. 2010 Oct;59(10):1401-9. doi: 10.1136/gut.2010.207423. Epub 2010 Jul 30. PMID 20675691
- [Derived] Morgan TR, Ghany MG, Kim HY, Snow KK, Shiffman ML, De Santo JL, Lee WM, Di Bisceglie AM, Bonkovsky HL, Dienstag JL, Morishima C, Lindsay KL, Lok AS; HALT-C Trial Group. Outcome of sustained virological responders with histologically advanced chronic hepatitis C. Hepatology. 2010 Sep;52(3):833-44. doi: 10.1002/hep.23744. PMID 20564351
- [Derived] Seeff LB, Everson GT, Morgan TR, Curto TM, Lee WM, Ghany MG, Shiffman ML, Fontana RJ, Di Bisceglie AM, Bonkovsky HL, Dienstag JL; HALT-C Trial Group. Complication rate of percutaneous liver biopsies among persons with advanced chronic liver disease in the HALT-C trial. Clin Gastroenterol Hepatol. 2010 Oct;8(10):877-83. doi: 10.1016/j.cgh.2010.03.025. Epub 2010 Apr 1. PMID 20362695
- [Derived] Fontana RJ, Sanyal AJ, Ghany MG, Lee WM, Reid AE, Naishadham D, Everson GT, Kahn JA, Di Bisceglie AM, Szabo G, Morgan TR, Everhart JE; HALT-C Trial Group. Factors that determine the development and progression of gastroesophageal varices in patients with chronic hepatitis C. Gastroenterology. 2010 Jun;138(7):2321-31, 2331.e1-2. doi: 10.1053/j.gastro.2010.02.058. Epub 2010 Mar 6. PMID 20211180
- [Derived] Snow KK, Bonkovsky HL, Fontana RJ, Kim HY, Sterling RK, Di Bisceglie AM, Morgan TR, Dienstag JL, Ghany MG; HALT-C Trial Group. Changes in quality of life and sexual health are associated with low-dose peginterferon therapy and disease progression in patients with chronic hepatitis C. Aliment Pharmacol Ther. 2010 Apr;31(7):719-34. doi: 10.1111/j.1365-2036.2010.04235.x. Epub 2010 Jan 12. PMID 20070284
- [Derived] Lok AS, Sterling RK, Everhart JE, Wright EC, Hoefs JC, Di Bisceglie AM, Morgan TR, Kim HY, Lee WM, Bonkovsky HL, Dienstag JL; HALT-C Trial Group. Des-gamma-carboxy prothrombin and alpha-fetoprotein as biomarkers for the early detection of hepatocellular carcinoma. Gastroenterology. 2010 Feb;138(2):493-502. doi: 10.1053/j.gastro.2009.10.031. Epub 2009 Oct 20. PMID 19852963
- [Derived] Ghany MG, Lok AS, Everhart JE, Everson GT, Lee WM, Curto TM, Wright EC, Stoddard AM, Sterling RK, Di Bisceglie AM, Bonkovsky HL, Morishima C, Morgan TR, Dienstag JL; HALT-C Trial Group. Predicting clinical and histologic outcomes based on standard laboratory tests in advanced chronic hepatitis C. Gastroenterology. 2010 Jan;138(1):136-46. doi: 10.1053/j.gastro.2009.09.007. Epub 2009 Sep 18. PMID 19766643
- [Derived] Shiffman ML, Morishima C, Dienstag JL, Lindsay KL, Hoefs JC, Lee WM, Wright EC, Naishadham D, Everson GT, Lok AS, Di Bisceglie AM, Bonkovsky HL, Ghany MG; HALT-C Trial Group. Effect of HCV RNA suppression during peginterferon alfa-2a maintenance therapy on clinical outcomes in the HALT-C trial. Gastroenterology. 2009 Dec;137(6):1986-94. doi: 10.1053/j.gastro.2009.08.067. Epub 2009 Sep 10. PMID 19747918
- [Derived] Freedman ND, Everhart JE, Lindsay KL, Ghany MG, Curto TM, Shiffman ML, Lee WM, Lok AS, Di Bisceglie AM, Bonkovsky HL, Hoefs JC, Dienstag JL, Morishima C, Abnet CC, Sinha R; HALT-C Trial Group. Coffee intake is associated with lower rates of liver disease progression in chronic hepatitis C. Hepatology. 2009 Nov;50(5):1360-9. doi: 10.1002/hep.23162. PMID 19676128
- [Derived] Everhart JE, Lok AS, Kim HY, Morgan TR, Lindsay KL, Chung RT, Bonkovsky HL, Ghany MG; HALT-C Trial Group. Weight-related effects on disease progression in the hepatitis C antiviral long-term treatment against cirrhosis trial. Gastroenterology. 2009 Aug;137(2):549-57. doi: 10.1053/j.gastro.2009.05.007. Epub 2009 May 13. PMID 19445938
- [Derived] Lok AS, Everhart JE, Chung RT, Kim HY, Everson GT, Hoefs JC, Greenson JK, Sterling RK, Lindsay KL, Lee WM, Di Bisceglie AM, Bonkovsky HL, Ghany MG, Morishima C; HALT-C Trial Group. Evolution of hepatic steatosis in patients with advanced hepatitis C: results from the hepatitis C antiviral long-term treatment against cirrhosis (HALT-C) trial. Hepatology. 2009 Jun;49(6):1828-37. doi: 10.1002/hep.22865. PMID 19291787
- [Derived] Lok AS, Seeff LB, Morgan TR, di Bisceglie AM, Sterling RK, Curto TM, Everson GT, Lindsay KL, Lee WM, Bonkovsky HL, Dienstag JL, Ghany MG, Morishima C, Goodman ZD; HALT-C Trial Group. Incidence of hepatocellular carcinoma and associated risk factors in hepatitis C-related advanced liver disease. Gastroenterology. 2009 Jan;136(1):138-48. doi: 10.1053/j.gastro.2008.09.014. Epub 2008 Sep 18. PMID 18848939
- [Derived] Lindsay KL, Morishima C, Wright EC, Dienstag JL, Shiffman ML, Everson GT, Lok AS, Bonkovsky HL, Lee WM, Morgan TR, Ghany MG; HALT-C Trial. Blunted cytopenias and weight loss: new correlates of virologic null response to re-treatment of chronic hepatitis C. Clin Gastroenterol Hepatol. 2008 Feb;6(2):234-41. doi: 10.1016/j.cgh.2007.11.020. PMID 18237873

RESULTS

PARTICIPANT FLOW:
Groups:
- Peginterferon Alfa-2a 90 mcg/Week: Treatment with Peginterferon alfa-2a 90 mcg administered once weekly for an additional 42 months
- Standard of Care Followup: Stop any peginterferon alfa-2a/ribavirin therapy and followed prospectively for an additional 42 months without treatment
Period: Overall Study
Arm/Group | Peginterferon Alfa-2a 90 mcg/Week | Standard of Care Followup
Started | 517 | 533
Completed | 447 (70 Withdrew or were lost to followup; 158 Discontinued peginterferon but were followed) | 452 (81 Withdrew or were lost to followup; 9 took peginterferon outside of protocol)
Not Completed | 70 | 81
Not completed — Withdrew or lost to follow-up | 70 | 81

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peginterferon Alfa-2a 90 mcg/Week | Standard of Care Followup | Total
Number analyzed (Participants) | 517 | 533 | 1050
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 489 | 511 | 1000
  >=65 years | 28 | 22 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (7.3) | 50.1 (7.0) | 50.6 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155 | 150 | 305
  Male | 362 | 383 | 745
Region of Enrollment [Number; unit: participants]
  United States | 517 | 533 | 1050

OUTCOME MEASURES:

1. Primary Outcome: Progression of Liver Disease as Indicated by Death, Hepatic Decompensation, Hepatocellular Carcinoma, or for Patients With Noncirrhotic Fibrosis at Baseline, an Increase in the Ishak Hepatic Fibrosis Score of 2 or More Points
Description: Progression of liver disease within 1400 days as indicated by death, hepatic decompensation (variceal hemorrhage; ascites; spontaneous bacterial peritonitis; hepatic encephalopathy), hepatocellular carcinoma, a Child-Turcotte-Pugh (CTP) score of 7 or more on two consecutive study visits (score range 5-15, higher score indicates greater decompensation), or for patients with noncirrhotic fibrosis at baseline, an increase in Ishak hepatic fibrosis score (range 0-6, higher score indicates greater fibrosis) of at least 2 points by assessment of a liver-biopsy specimen obtained during the study
Time Frame: 1400 days (3.85 years) post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Peginterferon Alfa-2a 90 mcg/Week | Standard of Care Followup
Number analyzed (Participants) | 517 | 533
Participants | 157 | 157

2. Primary Outcome: Increase in Ishak Fibrosis Score by 2 Points or More at 2 or 4 Year Biopsies
Description: For patients with noncirrhotic fibrosis at baseline, an increase in Ishak hepatic fibrosis score (range 0-6, higher score indicates greater fibrosis) of at least 2 points by assessment of a liver-biopsy specimen obtained during the study (collected at Year 2 and Year 4 biopsies, 1.5 and 3.5 years after randomization)
Time Frame: 1400 days (3.85 years) post randomization
Population: Patients with Ishak fibrosis score <5 at baseline and at least one follow-up biopsy
Measure: Count of Participants; unit: Participants
Arm/Group | Peginterferon Alfa-2a 90 mcg/Week | Standard of Care Followup
Number analyzed (Participants) | 273 | 274
Participants | 71 | 81

3. Primary Outcome: Death From Any Cause
Time Frame: 1400 days (3.85 years) post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Peginterferon Alfa-2a 90 mcg/Week | Standard of Care Followup
Number analyzed (Participants) | 517 | 533
Participants | 31 | 22

4. Primary Outcome: Development of Hepatocellular Carcinoma (HCC)
Description: A diagnosis of development of hepatocellular carcinoma (HCC) was based on either
  1. Histology showing HCC (from a biopsy, surgery, or autopsy) or
  2. A new hepatic defect on imaging with an alpha-fetoproteion (AFP) level rising to > 1,000 ng/ml.
Time Frame: 1400 days (3.85 years) post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Peginterferon Alfa-2a 90 mcg/Week | Standard of Care Followup
Number analyzed (Participants) | 517 | 533
Participants | 13 | 16

5. Primary Outcome: Child-Turcotte-Pugh (CTP) Score of 7 or Higher at Two Consecutive Study Visits
Description: Child-Turcotte-Pugh (CTP) score of 7 or more on two consecutive study visits (score range 5-15, higher score indicates greater hepatic decompensation)
Time Frame: 1400 days (3.85 years) post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Peginterferon Alfa-2a 90 mcg/Week | Standard of Care Followup
Number analyzed (Participants) | 517 | 533
Participants | 57 | 52

6. Primary Outcome: Variceal Hemorrhage
Description: A gastrointestinal hemorrhage which is believed by the investigator to be due to bleeding esophageal or gastric varices. In general, an endoscopy will have been performed and will have revealed either direct evidence of variceal bleeding (bleeding varix, red wale sign) or historical evidence for significant upper gastro-intestinal bleeding plus upper endoscopy revealing moderate varices and no other site of bleeding is identified
Time Frame: 1400 days (3.85 years) post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Peginterferon Alfa-2a 90 mcg/Week | Standard of Care Followup
Number analyzed (Participants) | 517 | 533
Participants | 5 | 11

7. Primary Outcome: Ascites
Description: Any abdominal fluid which is:
  1. Mild, moderate or marked on ultrasound; or
  2. Progressive on serial physical examinations; or
  3. Requires diuretic therapy. To meet the definition of ascites, abdominal fluid that is "mild" ("barely detectable") on physical examination requires ultrasound confirmation that is "mild", "moderate" or "marked" ascites. Ultrasound reports of minimal fluid around the liver do not meet the definition.
Time Frame: 1400 days (3.85 years) post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Peginterferon Alfa-2a 90 mcg/Week | Standard of Care Followup
Number analyzed (Participants) | 517 | 533
Participants | 32 | 27

8. Primary Outcome: Spontaneous Bacterial Peritonitis
Description: Any episode of spontaneous ascitic infection diagnosed on the basis of elevated neutrophil count (> 250/ml) in paracentesis fluid or positive bacterial cultures and clinical diagnosis in the absence of white blood cell (WBC) availability.
Time Frame: 1400 days (3.85 years) post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Peginterferon Alfa-2a 90 mcg/Week | Standard of Care Followup
Number analyzed (Participants) | 517 | 533
Participants | 3 | 3

9. Primary Outcome: Hepatic Encephalopathy
Description: Any mental status alteration which is deemed by the investigator to be due to portosystemic encephalopathy, whether occurring during a provoked episode (GI bleeding, diuretics, usual sedative doses), or spontaneously (without apparent cause).
Time Frame: 1400 days (3.85 years) post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Peginterferon Alfa-2a 90 mcg/Week | Standard of Care Followup
Number analyzed (Participants) | 517 | 533
Participants | 15 | 22

10. Secondary Outcome: Serious Adverse Events
Description: A serious adverse event (SAE) is an untoward medical occurrence that results in any of the following:
  1. Death
  2. Is life threatening (risk of death at the time of the event)
  3. Requires in-patient hospitalization or prolongation of existing hospitalization
  4. Results in persistent or significant disability/incapacity
  5. Congenital abnormality or birth defect
  Trial outcomes (except death) were not considered serious adverse events.
Time Frame: 1400 days (3.85 years) post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Peginterferon Alfa-2a 90 mcg/Week | Standard of Care Followup
Number analyzed (Participants) | 517 | 533
Participants | 175 | 155

11. Secondary Outcome: Changes in Fibrosis From Baseline at Year 2 or Year 4 Biopsy.
Description: Change in Ishak hepatic fibrosis score (range 0-6, higher score indicates greater fibrosis) by assessment of a liver-biopsy specimen obtained during the study (collected at baseline, Year 2 and Year 4 biopsies, 1.5 and 3.5 years after randomization)
Time Frame: 1400 days (3.85 years) post randomization
Population: Numbers of participants at 1.5 and 3.5 years are the number with biopsies at those time points
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peginterferon Alfa-2a 90 mcg/Week | Standard of Care Followup
Number analyzed (Participants) | 430 | 429
units on a scale
  1.5 years | -0.07 (1.27) | -0.09 (1.27)
  3.5 years: number analyzed (Participants) | 349 | 350
  3.5 years | 0.12 (1.36) | 0.12 (1.43)

12. Secondary Outcome: Presumed Hepatocellular Carcinoma (HCC)
Description: Presumed HCC was considered when histology was not available and alpha-fetoprotein (AFP) is <1000 ng/ml, if:
  1. A new hepatic lesion was shown on ultrasound and 1 additional imaging showed a hepatic lesion with characteristics of HCC.
  2. AFP> upper limit of normal (ULN) and 2 imaging studies showed a hepatic lesion with characteristics of HCC.
  3. A progressively enlarging hepatic lesion starting as a new defect resulting in patient death.
  4. A new hepatic defect with at least 1 characteristic scan and:
     1. Increase in size over time or
     2. Increasing AFP rising to a level of >200 ng/ml
Time Frame: 1400 days (3.85 years) post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Peginterferon Alfa-2a 90 mcg/Week | Standard of Care Followup
Number analyzed (Participants) | 517 | 533
Participants | 10 | 9

13. Secondary Outcome: SF-36 Vitality Summary Score
Description: Change from baseline to years 0.5, 1.5, 2.5, and 3.5 in Short Form Health Survey (SF-36) Vitality summary score. The SF-36 Vitality summary score is the sum of 4 individual scores. It is scaled from 0 to 100 with a score of 0 equivalent to maximum disability and a score of 100 equivalent to no disability. A negative value indicates a decrease in quality of life from baseline.
Time Frame: 0.5, 1.5, 2.5, and 3.5 years after randomization
Population: At each visit the analysis population is the number who completed the questionaire
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peginterferon Alfa-2a 90 mcg/Week | Standard of Care Followup
Number analyzed (Participants) | 517 | 533
units on a scale
  0.5 years: number analyzed (Participants) | 487 | 492
  0.5 years | -6.05 (20.5) | -1.61 (19.5)
  1.5 years: number analyzed (Participants) | 468 | 471
  1.5 years | -6.40 (20.31) | -3.24 (20.34)
  2.5 years: number analyzed (Participants) | 436 | 430
  2.5 years | -5.68 (21.71) | -2.97 (19.73)
  3.5 years: number analyzed (Participants) | 226 | 214
  3.5 years | -6.69 (19.83) | -3.27 (23.3)

14. Secondary Outcome: SF-36 Physical Function Summary Score
Description: Change from baseline to years 0.5, 1.5, 2.5, and 3.5 in Short Form Health Survey (SF-36) Physical Function summary score. The SF-36 Physical Function summary score is the sum of 10 individual scores. It is scaled from 0 to 100 with a score of 0 equivalent to maximum disability and a score of 100 equivalent to no disability. A negative value indicates a decrease in quality of life from baseline.
Time Frame: 0.5, 1.5, 2.5, and 3.5 years after randomization
Population: At each visit the analysis population is the number who completed the questionaire
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peginterferon Alfa-2a 90 mcg/Week | Standard of Care Followup
Number analyzed (Participants) | 517 | 533
units on a scale
  0.5 years: number analyzed (Participants) | 483 | 485
  0.5 years | -1.64 (8.66) | -0.97 (8.52)
  1.5 years: number analyzed (Participants) | 460 | 467
  1.5 years | -2.41 (9.10) | -1.63 (9.29)
  2.5 years: number analyzed (Participants) | 434 | 426
  2.5 years | -1.99 (9.87) | -1.68 (9.23)
  3.5 years: number analyzed (Participants) | 223 | 213
  3.5 years | -3.80 (9.56) | -1.66 (9.10)

15. Secondary Outcome: SF-36 Mental Health Summary Score
Description: Change from baseline to years 0.5, 1.5, 2.5, and 3.5 in Short Form Health Survey (SF-36) Mental Health summary score. The SF-36 Mental Health summary score is the sum of 5 individual scores. It is scaled from 0 to 100 with a score of 0 equivalent to maximum disability and a score of 100 equivalent to no disability. A negative value indicates a decrease in quality of life from baseline.
Time Frame: 0.5, 1.5, 2.5, and 3.5 years after randomization
Population: At each visit the analysis population is the number who completed the questionaire
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peginterferon Alfa-2a 90 mcg/Week | Standard of Care Followup
Number analyzed (Participants) | 517 | 533
units on a scale
  0.5 years: number analyzed (Participants) | 483 | 485
  0.5 years | -2.62 (9.58) | -1.08 (9.73)
  1.5 years: number analyzed (Participants) | 460 | 467
  1.5 years | -2.22 (9.68) | -1.67 (9.57)
  2.5 years: number analyzed (Participants) | 434 | 426
  2.5 years | -2.65 (10.17) | -2.15 (10.00)
  3.5 years: number analyzed (Participants) | 223 | 213
  3.5 years | -2.84 (9.56) | -1.85 (10.88)

ADVERSE EVENTS:
Time Frame: Within 1400 days (3.83 years) after randomization
Description: In the treatment group, 3991 adverse events occurred among 486 patients, as compared with 3129 adverse events among 492 patients in the control group; 330 patients had at least one serious adverse event.
Arm/Group | Peginterferon Alfa-2a 90 mcg/Week | Standard of Care Followup
Serious Adverse Events (participants affected / at risk) | 175/517 | 155/533
Other Adverse Events (participants affected / at risk) | 486/517 | 492/533
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peginterferon Alfa-2a 90 mcg/Week (N=517) | Standard of Care Followup (N=533)
Anemia (Blood and lymphatic system disorders) | 3 | 5
Thrombocytopenia or pancytopenia (Blood and lymphatic system disorders) | 4 | 0
Atherosclerotic disease (Cardiac disorders) | 16 | 9
Arrhythmia (Cardiac disorders) | 3 | 9
Other cardiovascular or circulatory event (Cardiac disorders) | 4 | 5
Nonvariceal gastrointestinal bleeding (Gastrointestinal disorders) | 4 | 9
Hernia or intestinal obstruction (Gastrointestinal disorders) | 5 | 3
Other digestive system event (Gastrointestinal disorders) | 11 | 15
Electrolyte, mineral, or water imbalance (Endocrine disorders) | 6 | 7
Diabetes and its complications (Endocrine disorders) | 1 | 2
Thyroid disease (Endocrine disorders) | 2 | 2
Renal or urinary diseases (Renal and urinary disorders) | 11 | 8
Gynecologic, menstrual, or sexual disorders (Reproductive system and breast disorders) | 2 | 5
Gallbladder disease (Hepatobiliary disorders) | 13 | 15
Other pancreatic or biliary disorders (Hepatobiliary disorders) | 7 | 5
Liver-disease events other than primary or secondary outcomes (Hepatobiliary disorders) | 1 | 1 — Liver-disease events not related to death or other study-related clinical primary or secondary outcomes of the trial
Mucocutaneous infection and infectious diseases (Infections and infestations) | 9 | 16
Respiratory tract infections and infectious diseases (Infections and infestations) | 19 | 11
Systemic infections and infectious diseases (Infections and infestations) | 10 | 4
Other infections and infectious diseases (Infections and infestations) | 15 | 19
Injury (Injury, poisoning and procedural complications) | 4 | 10
Drug reaction (Injury, poisoning and procedural complications) | 4 | 2
Liver-biopsy complication (Injury, poisoning and procedural complications) | 8 | 11
Musculoskelatal surgery (Musculoskeletal and connective tissue disorders) | 25 | 21
Arthritis or back pain (Musculoskeletal and connective tissue disorders) | 9 | 6
Malignant neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 10
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Cerebral aneurysm, infarct, or stroke (Nervous system disorders) | 3 | 4
Other neurologic event (Nervous system disorders) | 3 | 2
Affective disorders or delirium (Psychiatric disorders) | 8 | 4
Suicidal ideation or attempt (Psychiatric disorders) | 4 | 4
Substance abuse (Psychiatric disorders) | 3 | 1
Respiratory disorders (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Benign skin and nail disorders (Skin and subcutaneous tissue disorders) | 0 | 2
Cardiovascular signs or symptoms (General disorders) | 10 | 6 — These clinical signs and symptoms are not associated with a specific diagnosis but are still classified as a serious adverse event.
Hepatobiliary signs or symptoms (General disorders) | 8 | 6 — These clinical signs and symptoms are not associated with a specific diagnosis but are still classified as a serious adverse event.
Neurologic signs or symptoms (General disorders) | 7 | 6 — These clinical signs and symptoms are not associated with a specific diagnosis but are still classified as a serious adverse event.
Digestive signs or symptoms (General disorders) | 4 | 3 — These clinical signs and symptoms are not associated with a specific diagnosis but are still classified as a serious adverse event.
Other general signs or symptoms (General disorders) | 4 | 8 — These clinical signs and symptoms are not associated with a specific diagnosis but are still classified as a serious adverse event.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Peginterferon Alfa-2a 90 mcg/Week (N=517) | Standard of Care Followup (N=533)
Anemia (Blood and lymphatic system disorders) | 26 | 11
Hypertension (Cardiac disorders) | 42 | 46
Diabetes (Endocrine disorders) | 33 | 56
Sexual dysfunction, impotence (Reproductive system and breast disorders) | 28 | 12
Cystitis, bladder infection (Infections and infestations) | 41 | 28
Pharyngitis (Infections and infestations) | 26 | 13
Pneumonia (Immune system disorders) | 27 | 23
Sinusitis (Infections and infestations) | 56 | 37
Upper respiratory infection (Infections and infestations) | 44 | 57
Arthralgia (Musculoskeletal and connective tissue disorders) | 136 | 119
Bursitis, tendonitis, enthesopathies (Musculoskeletal and connective tissue disorders) | 14 | 27
Limb pain (Musculoskeletal and connective tissue disorders) | 36 | 38
Muscle spasm (Musculoskeletal and connective tissue disorders) | 52 | 32
Muscle/back aches or pain (Musculoskeletal and connective tissue disorders) | 145 | 124
Anxiety (Psychiatric disorders) | 27 | 29
Depression (Psychiatric disorders) | 93 | 89
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 27 | 24
Chest pain (General disorders) | 42 | 39
Diarrhea, loose stool (General disorders) | 48 | 39
Nausea (General disorders) | 52 | 34
Abdominal pain (Hepatobiliary disorders) | 136 | 134
Dizziness, vertigo, light-headedness (General disorders) | 42 | 31
Headache (General disorders) | 77 | 44
Insomnia, sleep disturbance (General disorders) | 92 | 54
Memory loss, confusion (General disorders) | 58 | 37
Tingling, numbness (General disorders) | 47 | 21
Nervousness, irritability (General disorders) | 62 | 23
Nonproductive cough (General disorders) | 34 | 22
Dyspnea (General disorders) | 26 | 18
Rash (General disorders) | 71 | 45
Body aches, chills, fever (General disorders) | 86 | 49
Fatigue, malaise, weakness (General disorders) | 141 | 121
Localized edema (General disorders) | 63 | 64
Pruritis (Skin and subcutaneous tissue disorders) | 93 | 70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No